CLINICAL TRIAL: NCT04097470
Title: A Randomized Phase II Multicenter Study to Assess the Tolerability and Efficacy of the Addition of Midostaurin to 10-day Decitabine Treatment in Unfit Adult Acute Myeloid Leukemia and High Risk Myelodysplasia Patients
Brief Title: Tolerability and Efficacy of Midostaurin to 10-day Decitabine in Unfit Adult AML and High Risk MDS Patients
Acronym: HO155
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOVON 155 AML; 2018-000047-31 (EudraCT Number); 2018-674 (Other: METc UMCG); NL64632.042.18 (Other: CCMO)
Record Dates: First submitted 2019-03-25; First posted 2019-09-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: AML/MDS
MeSH Terms: interventions — Decitabine; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Decitabine (Active Comparator): Cycles 1-3: Decitabine 10-day; depending on day +28 bone marrow (BM) blasts after the previous cycle, next cycle consists of either 5-day (BM blasts < 5%) or 10-day (BM blasts ≥5%) decitabine. Cycles 4 and beyond: 5-day decitabine (in cycles of 4-8 weeks); continuation of these cycles until progression.
  Dosage for Decitabine 20 mg/m2 i.v.
  Interventions: Drug: Decitabine
- Arm B: Decitabine and Midostaurin (Experimental): Cycle 1:Decitabine; 10-day schedule (start day +1) + midostaurin (start day +11). Midostaurin is given until 2 days before start next cycle of decitabine. Cycles 2-3: Decitabine 5 or 10-day schedule; depending on day +28 bone marrow blasts of the previous cycle, next cycle consist of either 5-day (BM blasts < 5%) or 10-day (BM blasts ≥5%) decitabine + midostaurin (daily, starting the day after the last dose of decitabine (i.e. day +6 or +11). Midostaurin is given until 2 days before start next cycle. Cycles 4 and beyond: 5-day decitabine (in cycles of 4-8 weeks) followed by midostaurin starting at day +6 until two days before start of next cycle of decitabine; continuation of these cycles until progression. Midostaurin is given until 2 days before start next cycle of decitabine.
  Dosage for Decitabine 20 mg/m2 i.v.
  Dosage for Midostaurin 50 mg b.i.d.
  Interventions: Drug: Decitabine; Drug: Midostaurin

INTERVENTIONS:
Drug: Decitabine — Decitabine dosage 20mg/m2 i.v.
  Other Names: Dacogen
Drug: Midostaurin — Midostaurin 50 mg b.i.d.
  Other Names: Rydapt
  Arms: Arm B: Decitabine and Midostaurin

SUMMARY:
The aim of this study is to investigate how safe and effective the addition of the new medicine midostaurin to decitabine is for the treatment of unfit acute myeloid leukemia (AML) and high-risk myelodysplasia (MDS) patients. Patients who are ineligible for intensive chemotherapy because of accompanying diseases may opt for gentler treatment. This does not produce a cure but serves to allow the quality of life to be acceptable for as long as possible. Decitabine is an example of a gentler treatment. It is effective against leukemia and has fewer side effects than intensive chemotherapy. Given in courses of 5 successive days, decitabine is registered for the treatment of AML. There is scientific research to suggest that decitabine is more effective and generally well tolerated when given in courses of 10 successive days. Therefore, treatment with 10-day courses of decitabine is the standard treatment in this scientific research. The aim is to investigate whether this standard treatment can be improved by adding a new product, midostaurin. Midostaurin is a medicine that is directed against a specific protein on leukaemia cells (FLT3).

DETAILED DESCRIPTION:
This trial aims to develop effective treatments for unfit (i.e. Hematopoietic cell transplantation co-morbidity index (HCT-CI) ≥ 3) in adult (≥ 18 yrs) AML patients, for whom current treatment strategies are highly unsatisfactory. Therefore new treatment modalities are introduced and evaluated in multiple parallel randomized phase II studies that will be conducted within the frame of a master protocol. The scheme of this new design consists of one arm with one of the currently considered best available treatments for unfit AML patients (i.e. 10-day decitabine). After a maximum of 3 10-day courses, or less in case of good response, treatment will be continued with 5-day decitabine courses. This treatment will be compared to investigational treatments in combination with decitabine.

The competitor of the 10-day decitabine schedule will be 10-day decitabine combined (sequential) with the tyrosine kinase inhibitor midostaurin (independent of the presence of FLT3 mutations). The rationale for midostaurin is: 1) single agent midostaurin has shown efficacy in both FLT3 wild type and mutant AML; 2) it has shown efficacy in a phase III randomized controlled trial when combined with intensive chemotherapy in FLT3-mutated AML (RATIFY study); 3) midostaurin has been successfully combined with hypomethylating agents (azacitidine and decitabine) and improved the response compared with historical response rates of these drugs, suggesting at least additive affects of midostaurin with hypomethylating agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients with:

  * a diagnosis of AML and related precursor neoplasms according to WHO 2016 classification (excluding acute promyelocytic leukemia) including secondary AML (after an antecedent hematological disease (e.g. MDS) and therapy-related AML, or
  * a diagnosis of myelodysplastic syndrome with excess of blasts (MDS) and International Prognostic Score System (IPSS) > 4.5
* Patients 18 years and older.
* Patients NOT eligible for standard chemotherapy, defined as hematopoietic cell transplantation comorbidity index (HCT-CI) ≥ 3.

or Patients NOT eligible for standard chemotherapy for other reasons (wish of patient).

* White blood cell (WBC) ≤ 30 x109/L (prior hydroxyurea allowed for a maximum of 5 days, stop 2 days before start decitabine treatment)
* Adequate renal and hepatic functions unless clearly disease related as indicated by the following laboratory values:

  * Serum creatinine ≤ 221.7 µmol/L (≤ 2.5 mg/dL ), unless considered AML-related
  * Serum bilirubin ≤ 2.5 x upper limit of normal (ULN), unless considered AML-related or due to Gilbert's syndrome
  * Alanine transaminase (ALT) ≤ 2.5 x ULN, unless considered AML-related
* WHO performance status 0, 1 or 2.
* Patient is willing and able to use adequate contraception during and until 5 months after the last protocol treatment.
* Written informed consent.
* Patient is capable of giving informed consent.

Exclusion Criteria:

* Acute promyelocytic leukemia.
* Acute leukemia's of ambiguous lineage according to WHO 2016
* Patient has symptomatic central nervous system (CNS) leukemia (NO routinely lumbar puncture required to investigate CNS involvement)
* Blast crisis of chronic myeloid leukemia.
* Diagnosis of any previous or concomitant malignancy is an exclusion criterion:
* except when the patient completed successfully treatment (chemotherapy and/or surgery and/or radiotherapy) with curative intent for this malignancy at least 6 months prior to randomization. OR
* except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix
* Patients previously treated for AML (any antileukemic therapy including investigational agents), a short treatment period ( ≤ 5 days) with Hydroxyurea is allowed
* Current concomitant chemotherapy, radiation therapy, or immunotherapy; other than hydroxyurea
* Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, pulmonary disease etc.)
* Cardiac dysfunction as defined by:

  * Myocardial infarction within the last 3 months of study entry, or
  * Reduced left ventricular function with an ejection fraction < 40% as measured by MUGA scan or echocardiogram or
  * Unstable angina or
  * New York Heart Association grade IV congestive heart failure or
  * Unstable cardiac arrhythmias.
* History of stroke or intracranial hemorrhage within 6 months prior to randomization.
* Patient has a history of human immunodeficiency virus or active infection with Hepatitis C or B.
* Patients known to be pregnant
* Patients with a history of non-compliance to medical regimens or who are considered unreliable with respect to compliance.
* Patients with any serious concomitant medical condition which could, in the opinion of the investigator, compromise participation in the study.
* Patients who have senile dementia, mental impairment or any other psychiatric disorder that prohibits the patient from understanding and giving informed consent.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative Complete Remission (CR) / CR with incomplete blood count (CRi) rate | 4-5 months
  Cumulative CR/CRi rate during 3 cycles

SECONDARY OUTCOMES:
Safety and tolerability of midostaurin determined by the type, frequency, severity and relationship of adverse events to study treatment | 5 years
  Safety and tolerability of midostaurin added to 10-day decitabine treatment for AML (type, frequency, severity and relationship of adverse events to study treatment).
Efficacy profile | 4-9 months
  The response rate after first three cycles together with the best response during three cycles and after 9 months will determinine the efficacy profile.
Event free survival (EFS) | 5 years
  The time from registration to induction failure, death or relapse whichever occurs first).
Overall survival (OS) | 5 years
  The time from the date of randomization to the date of death, whatever the cause. Patients still alive at the date last contact will be censored.
Hospital stay duration | 4-5 months
  Days of staying in hospital during 3 cycles.
Transfusion need | 4-5 months
  Number of participants with transfusion needs during 3 cycles.
Prognostic value of MRD | 9 months and at relapse
  Assessment of the prognostic value of Minimal Residual Disease (MRD) by flowcytometry or PCR
Predictive value of gene mutations | 5 years
  Assessment of the predictive value of gene mutations by exploratory analysis
Prognostic value of baseline physical conditions as measured by the short physical performance battery | 5 years
  Assessment of the prognostic value of baseline physical and functional conditions using a comprehensive geriatric assessment tool, short physical performance battery (SPPB), on treatment outcome. Total scores (range 0 to 12) will be used to determine physical performance.
Prognostic value of baseline functional conditions as measured by the activities of daily living | 5 years
  Assessment of the prognostic value of baseline functional conditions using a comprehensive geriatric assessment tool, activities of daily living (ADL), on treatment outcome. Total points (range 0 to 6) will be used to determine functional condition.

CONTACTS AND LOCATIONS:
Overall Officials: Gerwin Huls, Prof, Principal Investigator — UMCG / HOVON
Locations (37):
- Belgium (3):
  - BE-Antwerpen-ZNASTUIVENBERG, Antwerp
  - BE-Haine-Saint-Paul-JOLIMONT, Haine-Saint-Paul
  - BE-Roeselare-AZDELTA, Roeselare
- DE-Magdeburg-OVGU, Magdeburg, Germany
- Netherlands (23):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam-OLVG, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Breda-AMPHIA, Breda
  - NL-Delft-RDGG, Delft
  - NL-Doetinchem-SLINGELAND, Doetinchem
  - NL-Dordrecht-ASZ, Dordrecht
  - NL-Ede-ZGV, Ede
  - NL-Eindhoven-CATHARINA, Eindhoven
  - NL-Eindhoven-MAXIMAMC, Eindhoven
  - NL-Enschede-MST, Enschede
  - NL-Groningen-UMCG, Groningen
  - NL-Leeuwarden-MCL, Leeuwarden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nieuwegein-ANTONIUS, Nieuwegein
  - NL-Nijmegen-CWZ, Nijmegen
  - NL-Nijmegen-RADBOUDUMC, Nijmegen
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Den Haag-HAGA, The Hague
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Zwolle-ISALA, Zwolle
- Switzerland (10):
  - CH-Aarau-KSA, Aarau
  - CH-Basel-USB, Basel
  - CH-Bellinzona-IOSI, Bellinzona
  - CH-Bern-INSEL, Bern
  - CH-Fribourg-HFR, Fribourg
  - CH-Geneve (14)-HCUGE, Geneva
  - CH-Lausanne-CHUV, Lausanne
  - CH-Luzern-LUKS, Lucerne
  - CH-St. Gallen-KSSG, Sankt Gallen
  - CH-Zürich-USZ, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HOVON website — http://www.hovon.nl